CLINICAL TRIAL: NCT06954467
Title: A Phase II, Open-label, Multi-center Study to Evaluate the Safety and Efficacy of JS207 Combined With JS007 as First-line Treatment for Advanced Hepatocellular Carcinoma（HCC）
Brief Title: JS207 Combined With JS007 as First-line Treatment for Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JS207-006-II-HCC
Record Dates: First submitted 2025-04-18; First posted 2025-05-01 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JS207 Combined with JS007-ArmA (Experimental)
  Interventions: Drug: JS207; Drug: JS007
- JS207 monotherapy-ArmB (Experimental)
  Interventions: Drug: JS207

INTERVENTIONS:
Drug: JS207 — 10 mg/kg q3W or adjust the dose (e.g. 15 mg/kg) based on accumulated data on the safety and efficacy of JS207 from clinical studies.
Drug: JS007 — Dose exploration stage: C1-C4, group 1:3 mg/kg, C1D1 once (single dose); Group 2:3 mg/kg, D1, Q6W; Group 3:1 mg/kg,D1, Q3W; ≥C5, 1 mg/kg, Q6W; Dose expansion stage: according to the group medication confirmed in the dose exploration stage.
  Arms: JS207 Combined with JS007-ArmA

SUMMARY:
This open-label, multicenter phase II study was designed to evaluate the safety and efficacy of JS207 alone or in combination with JS007 as first-line treatment in subjects with advanced HCC.

The subjects were all subjects with unresectable, locally advanced, recurrent, or metastatic HCC who had not received previous systemic therapy. Planned to enroll 43 to 72 subjects.The study was divided into two stages, dose exploration stage (3-12 cases) and random expansion stage (40-60 cases).After the dose exploration phase, a dose group was selected to enter the randomized expansion phase based on comprehensive discussion and evaluation of DLT, AE, dose adjustment, PK parameters and preliminary efficacy results in each dose group.

DETAILED DESCRIPTION:
This open-label, multicenter phase II study was designed to evaluate the safety and efficacy of JS207 alone or in combination with JS007 as first-line treatment in subjects with advanced HCC.

The subjects were all subjects with unresectable, locally advanced, recurrent, or metastatic HCC who had not received previous systemic therapy. Planned to enroll 43 to 72 subjects.The study was divided into two stages, namely dose exploration stage (3-12 cases) and random expansion stage (40-60 cases).Dose-finding phase: This phase was designed to initially evaluate the tolerability and safety of JS207 combined with JS007 in patients with advanced HCC, and to determine the expansion dose. JS207 was administered at a fixed dose of 10 mg/kg every 3 weeks (Q3W). A Bayesian optimal interval (BOIN) design was used to explore the dose and frequency of JS007 administration (every 3-week treatment cycle, with a DLT observation period of 21±3 days after the first dose). For subjects who received the initial dose of dose 1 (a single dose of 3 mg/kg, 1 mg/kg every 6 weeks starting cycle 5 [Q6W]), the results were according to the BOIN design: if the dose was judged to be increased, dose 2 (3 mg/kg Q6W, 1 mg/kg Q6W starting cycle 5) was used for subsequent subjects. Dose 3 (1 mg/kg Q3W, followed by 1 mg/kg Q6W from cycle 5) was used for subsequent subjects if dose reduction or maintenance was judged. Dose 2 or dose 3 was similarly explored using the BOIN design.After the dose exploration phase, a dose group was selected to enter the randomized expansion phase based on comprehensive discussion and evaluation of DLT, AE, dose adjustment, PK parameters and preliminary efficacy results in each dose group.

Randomized expansion phase: This phase was designed to initially evaluate the efficacy of JS207 alone or in combination with JS007 in the first-line treatment of subjects with advanced HCC, as well as to further evaluate their safety. The randomized expansion phase planned to enroll approximately 40 to 60 subjects who would be randomly assigned in A 1:1 ratio to receive JS207 plus JS007 (cohort A) or JS207 alone (cohort B). Randomization stratification factor: baseline AFP level (<400ng/mL vs. ≥400ng/mL).Dose reductions or increases in JS207 and JS007 were not allowed during the study period, and drug interruptions or discontinuation were allowed. Neither JS207 nor JS007 was given for a maximum of 2 years. When a study drug was discontinued for any reason, the other study drugs could be continued.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate and sign a written informed consent form.
2. Age ≥ 18 years, male or female.
3. Patients with histologically/cytologically confirmed HCC or Hepatic cirrhosis meeting the criteria of the American Association for the Study of Liver Diseases (AASLD) can be enrolled.
4. HCC classified as Barcelona Clinic Liver Cancer (BCLC) stage B (intermediate stage) or stage C (advanced stage), or stage IIa/IIb or IIIa/IIIb as defined by the Primary Liver Cancer Diagnosis and Treatment Guidelines (2024 Edition), prior to lymph node clearance, and deemed unsuitable for surgical and/or local treatment.
5. No systemic therapy for HCC prior to study entry (mainly including systemic chemotherapy, targeted therapy, immunotherapy, etc.; adjuvant/neoadjuvant administration of small molecule anti-angiogenic drugs, such as lenvatinib, sorafenib, and donafenib, is allowed, but the last dose of these drugs must be administered ≥90 days prior to the first dose of the study drug).
6. Having ≥1 measurable lesion according to RECIST v1.1. Requirement: The selected target lesion had not been subjected to local therapy previously, or the selected target lesion was located in the area of previous local therapy, but later determined to be progressed through imaging examination according to RECIST v1.1.
7. Child-Pugh liver function class A or B ≤ 7 without history of Hepatic encephalopathy.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0-1.
9. Life expectancy ≥12 weeks.
10. Major organ function meets the following requirements, without transfusion, hematopoietic stimulating factors (including G-CSF, GM-CSF, EPO and TPO, etc.) or human Albumin preparations within 14 days prior to screening:
11. Females of childbearing potential and males whose partners are of childbearing age are required to use highly effective contraceptive measures during the trial and for at least 6 months after the last dose (Appendix 5). Female patients of childbearing potential must have a negative serum HCG test within 7 days before study entry and must be non-lactating.

Exclusion Criteria:

Participants who meet any of the following criteria should be excluded from this study:

1. Received major surgery (requiring general anesthesia and >24 hours of hospitalization, excluding diagnostic biopsy), live vaccination, or investigational drug treatment within 4 weeks prior to the first dose, or received palliative radiotherapy for localized bone/brain lesions within 2 weeks prior to the first dose.
2. Patients who are receiving chronic systemic corticosteroid therapy (daily dose >10 mg prednisone or other glucocorticoid with the same effect) or other immunosuppression therapy within 7 days prior to the first dose.
3. Hepatic tumor burden > 50% of total hepatic volume at screening.
4. Invasion of portal vein main trunk (Vp4) by cancer thrombus (more than 1/2 of lumen) as confirmed by CT/MRI examination.
5. Presence of metastases to central nervous system of HCC; MRI scan of brain and/or spine is required to rule out the possibility when it is suspected.
6. Toxicity induced by previous treatment (except for alopecia and Neuropathy peripheral) has not recovered to ≤ grade 1 (NCI-CTCAE v5.0).
7. Severe infection during the screening period, including but not limited to hospitalization for infection, bacteraemia or severe pneumonia complications, oral or intravenous administration of therapeutic antibiotics for ≥7 days within 14 days prior to the first dose (patients receiving prophylactic antibiotics can be enrolled), fever ≥38.5°C of unknown origin within 7 days prior to the first dose or white blood cell count >15×109/L at baseline.
8. Uncontrolled pericardial effusion, uncontrolled pleural effusion, or clinically evident moderate or severe peritoneal effusion during screening period is defined as meeting the following criteria: having clinical symptoms and detectable pericardial, pleural, and peritoneal effusion on physical examination; or pleural and peritoneal effusion requiring puncture and aspiration and/or intracavitary drug administration for treatment.
9. Grade ≥3 (NCI-CTCAE v5.0) gastrointestinal or non-gastrointestinal fistula during screening period.
10. Existence of severe unhealed wounds, active ulcer and Therapy naive fracture at screening period.
11. Severe cardiovascular diseases.
12. History of haemorrhage of digestive tract within 6 months prior to the first dose, or clear haemorrhagic diathesis (including high-risk severe esophageal-gastric varicose vein, local active digestive tract ulcer lesions, and persistent faecal occult blood positive; if faecal occult blood positive at baseline, it can be rechecked; if still positive after recheck, upper gastrointestinal endoscopy is required; if endoscopy indicates severe esophageal-gastric varicose vein or the investigator judges that there is a clear risk of bleeding, then the subject cannot be enrolled).
13. Evidence of other haemorrhagic diathesis or significant coagulopathy.
14. History of intestinal obstruction and/or clinical signs or symptoms of gastrointestinal tract obstruction within 6 months prior to the first dose, including incomplete obstruction associated with pre-existing diseases requiring routine parenteral hydration, parenteral nutrition, or enteral feeding (patients who received definite [surgical] treatment prior to the first dose to resolve the obstruction symptoms were allowed to be enrolled).
15. Active autoimmune disorders requiring systemic treatment within 2 years prior to the first dose; however, replacement therapy (e.g., Thyroxine, Insulin, or physiological replacement of corticosteroids for adrenal or Pituitary insufficiency) will not be considered as systemic treatment and is allowed.
16. Having had neoplasm malignant (except HCC) within 5 years prior to the first dose, including mixed type of liver cancer; however, localized tumors that have been cured, including Carcinoma cervix in situ, Basal cell carcinoma, and Carcinoma in situ of prostate, etc.
17. History of interstitial lung disease or noninfectious pneumonitis, unless caused by local radiotherapy.
18. Patients with active tuberculosis or who have received anti-tuberculosis therapy within one year prior to the first dose.
19. HBV and/or HCV infection: a) HBsAg (+) and/or HBcAb (+), and HBV DNA > 1000 IU/mL (if the lower limit of the minimum measurable value of the local center is higher than 1000 IU/mL, enrollment will be decided according to the specific circumstances after discussion with the sponsor; the patient must continue to receive the original anti-HBV therapy throughout the study, or start the entecavir or tenofovir throughout the study after screening); b) positive HCV Antibody and HCV RNA > upper limit of normal; c) co-infection with hepatitis B and C.
20. Known history of human immunodeficiency virus (HIV) infection, prior allogeneic stem cell or Solid organ transplant, or other Immunodeficiency.
21. Known severe allergy to any Monoclonal antibodies.
22. Other factors that may affect the study results or cause the study to be terminated prematurely, as judged by the investigator, such as alcoholism, Drug of Abuse, other serious diseases (including mental disorders), need for concomitant treatment, serious Laboratory test abnormal, and family or social factors that may affect the patient's safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
AE | up to 27 mouths
  All adverse events, regardless of relationship to the study drug, were reported from the time the study drug was started until 90 days after the last dose or the subject started a new antineoplastic therapy, whichever occurred first.
SAE | up to 27 mouths
  Only those resulting from interventions required by the protocol were reported from the time of ICF signing until the first dose. All were reported from the time of the first dose until 90 days after the last dose or initiation of a new antineoplastic therapy, after which, those considered to be related to previous study treatment were reported.
DLT | up to 24 days after the first dose
  Dose-limiting toxicity
ORR | up to 27 mouths
  Objective remission rate

SECONDARY OUTCOMES:
PFS | up to 27 mouths
  Progression free survival
DCR | up to 27 mouths
  Disease control rate
DOR | up to 27 mouths
  Duration of response
OS | up to 27 mouths
  Overall survival
The trough concentrations（PK） | up to 27 mouths
  To characterize the trough concentrations of JS207 and JS007
Antidrug antibodies（ADA） | up to 27 mouths
  To characterize antidrug antibodies of JS207 and JS007
Neutralizing antibody（Nab） | up to 27 mouths
  To characterize neutralizing antibody of JS207 and JS007

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - The First Affiliated Hospital of USTC, Hefei, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Zhongshan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine City:Shanghai, Shanghai, Shanghai Municipality
  - Shanghai East Hospital,School of Medicine, Tongji University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No